CLINICAL TRIAL: NCT02897778
Title: A Phase 1 Cardiac Safety Study of Entinostat in Men and Women With Advanced Solid Tumors
Brief Title: Cardiac Safety Study of Entinostat in Men and Women With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNDX-275-0140
Record Dates: First submitted 2016-08-20; First posted 2016-09-13 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Digestive System Neoplasms; Endocrine Gland Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Breast Neoplasms; Breast Diseases; Renal Neoplasm; Solid Tumors
Keywords: entinostat; solid tumor; Histone Deacetylase Inhibitors
MeSH Terms: conditions — Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Digestive System Neoplasms; Endocrine Gland Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Breast Neoplasms; Breast Diseases; Kidney Neoplasms | interventions — entinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entinostat (Active Comparator): Participants received a single oral supratherapeutic dose of 15 mg entinostat under fasted conditions.
  Interventions: Drug: Entinostat
- Placebo (Placebo Comparator): Participants received a single dose of placebo-matching entinostat under fasted conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Entinostat — Single, supratherapeutic dose of entinostat given orally.
  Other Names: SNDX-275; MS-275
  Arms: Entinostat
Drug: Placebo — Single dose of placebo-matching entinostat (containing inactive ingredients matching the appearance of the active product).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of entinostat on heart rate and other electrocardiogram (ECG) parameters. This study will also evaluate the safety and tolerability of entinostat, as well as pharmacokinetic and pharmacodynamic parameters.

DETAILED DESCRIPTION:
This is a single center, randomized, placebo-controlled, single dosing schedule, double-blinded study to evaluate the effect of entinostat as compared to placebo on the electrical activity of the heart in patients with advanced solid tumors. Thirty patients will be randomized in a 1:1 ratio to receive either entinostat or placebo. Study treatment will be blinded to patients and the Investigator. ECG analysts will be blinded to the patient, visit, and treatment allocation. Patients will be on study up to 30 days following study drug administration. Total study duration is expected to be 9 months. After completing this study and at the discretion of the Investigator, patients may elect to enroll into a separate continuation study (SNDX-275-0141).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of a solid tumor malignancy that is not responsive to standard therapy(ies) or for which there is no approved therapy
* Patients must have acceptable laboratory requirements
* Left ventricular ejection fraction as measured by echocardiogram or multiple-gated acquisition scan that is above the institutional lower level of normal or greater than 50%
* Has experienced resolution of toxic effect(s) of the most recent prior chemotherapy and/or prior surgical and radiation treatment
* Must be able to understand and give written informed consent and comply with study procedures

Exclusion Criteria:

* If the patient has brain metastasis, they must have stable neurologic status without the use of steroids or on a stable or decreasing dose of steroids
* Presence of clinically significant gastrointestinal abnormalities that may affect the absorption of study treatments
* A medical condition that precludes adequate study treatment compliance or assessment, or increases patient risk in the opinion of the Investigator
* Patient has a concomitant cardiovascular issue that precludes adequate study treatment compliance or increases patient risk
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study
* Prior anti-cancer monoclonal antibody within 4 weeks prior to baseline
* Currently enrolled in another investigational study
* Has disease that is suitable for approved therapy administered with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Heart Rate (HR) | Baseline (pre-dose) through 24 hours post-dose
  Heart rate measured in beats per minute (bpm).
Change from Baseline in Electrocardiogram Procedures | Baseline (pre-dose) through 24 hours post-dose
  Change from baseline in QT interval corrected for heart rate (Qtc), PR interval (PR) and QRS complex (QRS).
Change from Baseline in T-Cell Morphology | Baseline (pre-dose) through 24 hours post-dose

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAES) and Serious Adverse Events (SAEs) | First dose through 30 days post-dose or through resolution of acute toxicities (Up to 31 days)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A TEAE is an AE that occurs after the first dose of study drug. A SAE is defined as any AE that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage.
Number of Participants with Clinically Significant Abnormalities in Laboratory Values Reported as a TEAE | Baseline (pre-dose) through 14 days post-dose or 30 day safety follow-up visit (if applicable)
  Standard safety laboratory tests included Chemistry, Hematology. Any hematologic or clinical chemistry abnormality considered by the investigator to be clinically significant was reported as a TEAE.
Change from Baseline in Vital Signs | Baseline (pre-dose) through 14 days post-dose or 30 day safety follow-up visit (if applicable)
  Vital signs included temperature, pulse, blood pressure, and respiration rate
Change from Baseline in ECG Values | Baseline ()pre-dose through 14 days post-dose or 30 day safety follow-up visit (if applicable)
  A 12-lead continuous ECG recording (via a Holter) was recorded on Day 1 for 25 hours. Safety ECGs were read and interpreted by the Investigator on-site for the purpose of safety monitoring and were transmitted electronically to the central ECG laboratory for clinical interpretation by a cardiologist
Change from Baseline in QTc | Pre-dose through 24 hours post-dose
Cmax (Maximum Plasma Concentration) of Entinostat when given as a Single Supratherapeutic Dose | Pre-dose and multiple time-points through 24 hours post-dose and 14 days post-dose
Tmax (Time of Maximum Plasma Concentration) of Entinostat when given as a Single Supratherapeutic Dose | Pre-dose and multiple time-points through 24 hours post-dose and 14 days post-dose
AUC0-24 (Area under the Plasma Concentration-time Curve from Time Zero to 24 hours) of Entinostat when given as a Single Supratherapeutic Dose | Pre-dose and multiple time-points through 24 hours post-dose and 14 days post-dose
AUC0-t (Area under the Plasma Concentration-time Curve from Time Zero to the Last Measurable Concentration) of Entinostat when given as a Single Supratherapeutic Dose | Pre-dose and multiple time-points through 24 hours post-dose and 14 days post-dose
AUC0-inf (Area under the Plasma Concentration-time Curve from 0-time Extrapolated to Infinity) of Entinostat when given as a Single Supratherapeutic Dose | Pre-dose and multiple time-points through 24 hours post-dose and 14 days post-dose
t1/2 (Elimination Half-life and Apparent Plasma Terminal Phase Elimination Rate Constant) of Entinostat when given as a Single Supratherapeutic Dose | Pre-dose and multiple time-points through 24 hours post-dose and 14 days post-dose
λz (Terminal Elimination Rate Constant) of Entinostat when given as a Single Supratherapeutic Dose | Pre-dose and multiple time-points through 24 hours post-dose and 14 days post-dose

OTHER OUTCOMES:
Changes in Immune Regulatory Cells after a Single Dose of Entinostat, when given at a Supratherapeutic Dose, Relative to Placebo Control | Pre-dose through 14 days post-dose
Variability and Changes in Protein Lysine Acetylation in Peripheral Blood Cells after a Single Dose of Entinostat, when given at a Supratherapeutic Dose and Examine the Underlying Biological Variation | Pre-dose through 14 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Michael Meyers, MD, PhD, Study Director — Syndax Pharmaceuticals
Locations (1):
- The START Center for Cancer Care, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be reviewed throughout the study by the sponsor, Contract Research Organization (CRO) assisting with Serious Adverse Event (SAE) management, and routine monitoring to safeguard the interests of trial patients and to assess the safety of the interventions administered during the trial.